CLINICAL TRIAL: NCT03675035
Title: A Prospective Study to Evaluate the Safety and Feasibility of an Endoluminal Suturing Device (Endominav2Mini) as an Aid for Pouch Reduction After Roux-And-Y-Gastric-Bypass Surgery
Brief Title: Endomina Post RYGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2017/360
Record Dates: First submitted 2018-08-27; First posted 2018-09-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endomina (Experimental): Reduction trough sutures of the gastro-jejunal anastomosis
  Interventions: Device: Endomina

INTERVENTIONS:
Device: Endomina — Reduction of the gastro-jejunal anastomosis through sutures

SUMMARY:
Surgery is the only effective treatment for morbid obesity and can be divided into restrictive surgeries (Lap Band and Sleeve gastrectomy), malabsorptive surgeries (Biliary pancreatic deviation and duodenal switch) or a combination of both (RYGBP).

This later technique is the most common and most effective surgical procedure performed worldwide and has been processed to be an effective treatment of morbid obesity and its complications, achieving excess weight loss of 65 to 80 % ; 1-2 years after surgery.1 However, after the initial weight loss induced by RYGBP; 50 % of patients regain some weight 2 and approximately 20 % of the patients will reach again a BMI of 35 at 10 years , defined as a failure rate.3 The reasons for weight regain are multiple but the most two potential contributing factors are related with the loss of the restrictive effect of the RYGBP by stretching of the gastric pouch and/or the gastrojejunal anastomosis (GJA), leading to increased satiety.

Surgical options available for treating weight regain after RYGBP include placement of adjustable gastric band, Redo of the anastomosis or Reconstruction of the pouch.4 These procedures are technically difficult especially in patients who had previous single or multiple surgical interventions leading to a morbidity of around 15 % and a mortality of 1 %; Which is twice the one of the original surgery. This justifies the interest in less invasive, peroral revisions that include injection of sclerosant or suturing the anastomosis using Endoluminal gastroplication device (EndoCinch; Bard) 5,6 They have been however of marginal effectiveness compared to the medical treatment may be because their effect is limited to the anastomosis and doesn't reduce the size of the stretched gastric pouch. StomaphyX (Endogastric Solutions, Redmond, WA) is another systems aiming to reduce the gastric pouch has proved initial efficacy but are disappointing on the long term by a lack of persistence of the plicators. 7, 8 Endomina (Endo Tools Therapeutics, Nivelles, Belgium) is CE mark robot driven device that may be attached to an endoscope inside the body and allows remote manipulation of the arms of devices during a peroral intervention. It offers the possibilities of making transoral surgical full thickness sutures and may allow performing, via a transoral route, an intervention combining anastomoses reduction and gastric pouch reduction. It might be an effective treatment option for patients regaining weight after RYGBP and having a stretched pouch and or anastomosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21-64 years;
2. BMI > 30 Kg/m2
3. Previous gastric bypass with limited results
4. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment , endoscopy, radiography, as well as laboratory investigations.
5. Must be able to understand and be willing to provide written informed consent.

Exclusion Criteria:

1. Achalasia and any other esophageal motility disorders
2. Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity.
3. Hypertension: uncontrolled hypertension during last 3 month
4. Severe renal, hepatic, pulmonary disease or cancer;
5. GIT stenosis or obstruction
6. Pregnancy or breastfeeding
7. Impending gastric surgery 60 days post intervention;
8. Currently participating in other study

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Adeverse Device Effect | 6 months post intervention
  Incidence of all adverse device effects

SECONDARY OUTCOMES:
Weight loss | 6 months post intervention
  difference between weight at intervention and after

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium